CLINICAL TRIAL: NCT06460623
Title: Comparative Effects of External Versus Rectal Coccygeal Mobilization on Symptom Severity, Disability & Quality of Life in Female With Coccydynia
Brief Title: Effect of Coccygeal Mobilization in Female With Coccydynia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0565
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Coccyx Disorder
Keywords: Coccyx,; Disability; Manipulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (external coccygeal mobilization+ stretching (Experimental): Patients lying prone received external mobilization as part of the study. Contact was made with the sacrospinous ligament and all soft tissue on the opposite side (e.g., if the coccyx was bent to the right, contact was made on the left). If the coccyx was bent to one side, the slack was taken up and stretched for five minutes. The manipulation group underwent two 5-minute sessions of external manipulation per week over a 5-week period.Burst TENS, which administers bursts of high-frequency pulses at a low frequency (less than 10 Hz), accompanied by a 10-minute application of a hot pack. Furthermore, muscle stretching, targeting the iliopsoas and piriformis, was conducted with a 30-second hold, comprising three sets of five repetitions per set.
  Interventions: Other: external mobilization
- internal coccygeal mobilization+ stretching (Active Comparator): . The investigator inserted the gloved and lubricated index finger of their right hand into the anal passage. The thumb of the investigator's other hand, also gloved but not lubricated, was placed on the dorsum of the coccyx to establish a good grasp between the two fingers. The technique involved distracting the coccyx along its long axis during the initial treatments,to correct alignment using controlled force in the coronal plane. The treatment consisted of two 5-minute sessions of external manipulation per week over a 5-week period.Burst TENS,less than 10 Hz accompanied by a 10-minute application of a hot pack. Furthermore, muscle stretching, targeting the iliopsoas and piriformis, was conducted with a 30-second hold, comprising three sets of five repetitions per set.
  Interventions: Other: rectal coccygeal mobilization

INTERVENTIONS:
Other: external mobilization — two 5-minute sessions of external manipulation per week over a 5-week period.
  Arms: (external coccygeal mobilization+ stretching
Other: rectal coccygeal mobilization — consisted of two 5-minute sessions of external manipulation per week over a 5-week period.
  Arms: internal coccygeal mobilization+ stretching

SUMMARY:
Aim of the study to evaluate the impact of mobilization on symptom severity, disability & quality of life in female with Coccydynia.

DETAILED DESCRIPTION:
In 2024, conducted a study to investigate the efficacy of combining manipulation and exercise in the treatment of coccydynia. Forty-six participants were split into two groups: an experimental group that received manipulation in addition to exercise, and a control group that received exercise only. As opposed to the exercise-only group, the manipulation group's members showed statistically significant reductions in pain, coccydynia symptoms, and disability scores at both the 6-month follow-up and immediately following treatment. In particular, there was a substantial drop in pain Visual Analog Scale scores from baseline to post-treatment (p < 0.001), and these scores persisted at the 6-month follow-up (p = 0.003). The manipulation group significantly reduced its Oswestry Disability Index scores from baseline to post-treatment (p < 0.001), and these scores continued to decline at the 6-month follow-up (p = 0.002). The Paris questionnaire scores for coccydynia symptoms also demonstrated a significant reduction in the manipulation group compared to the exercise-only group (p = 0.007). These results imply that for patients with persistent coccydynia, a brief course of intrarectal manipulation combined with exercise can significantly reduce pain and symptoms.

In 2023, conducted a single-blind randomized controlled trial study to evaluate the efficacy of adding kinesiotaping versus pelvic floor exercise to conventional therapy in the management of post-colonoscopy coccydynia. Forty-two participants, aged 25-45 years, were randomly assigned to: the conventional therapy group (CT) receiving Piriformis and Iliopsoas muscle stretching exercise, clamshell exercise, and seat cushioning; the CT plus kinesiotaping group (CT-KT) receiving additional kinesiotaping; or the CT plus pelvic floor exercise (PFE) group (CT-PFE) executing additional PFE. This study concluded thst CT-KT is more effective than CT-PFE in reducing pain associated with coccydynia post-colonoscopy, but there is no difference in their effects on functional disability. CT-KT is therefore recommended as an alternative treatment option for post-colonoscopy coccydynia.

In 2023 looked into the effects of a multimodal therapy approach on postpartum coccydynia in their randomized control experiment. 56 females, aged 25-35, with a VAS score ≥ 6 and more than two childbirths, were randomized into two groups: the control group (n = 28) and the intervention group (n = 28). Heat therapy, piriformis and iliopsoas muscle stretching, and coccyx and sacroiliac joint mobilization were administered to the intervention group. Comparing the treated group to the controls, the results showed substantial improvements (p<0.05) in pain intensity (VAS), tenderness (algometer), and pain-free sitting duration. Interestingly, after treatment, the intervention group's VAS ratings dropped from 6.87±2.07 to 3.9±1.37, while the controls' values went from 6.87±1.9 (pre-study) to 6.2±1.8 (post-study). This study offers insights into a helpful treatment plan for pain reduction and recovery, indicating that stretching, joint mobilization, and NSAIDs work well together to address postpartum Coccydynia.

In 2023,undertook a quality improvement (QI) study to assess the feasibility, acceptability, and therapeutic outcomes of transrectal osteopathic manipulative treatment (OMT) for persistent coccydynia in a primary care context. The study treated and evaluated 16 patients with chronic coccydynia in a primary care outpatient clinic using transrectal OMT, which included myofascial release and balanced ligamentous tension, as well as active patient movement of the head and neck. The study indicated that all 16 patients agreed to the OMT intervention, with six additionally receiving extra procedural therapy. Among the ten patients who only underwent OMT, post-treatment scores immediately after one procedure (acute model) improved significantly as compared to pretreatment levels.The mean pain scores on a 0-10 numerical rating scale (NRS) for coccydynia were reduced from 6.8 ± 1.2 before treatment to 3.2 ± 1.5 immediately after treatment. Five patients' pain levels at different intervals showed significant improvement, with a mean drop to 2.4 ± 1.6. The study indicated that transrectal OMT is a realistic and acceptable treatment option for coccydynia, with patients reporting satisfaction and improvement.

In 2022, conducted a prospective randomized studies to eevaluate the The Efficacy of Extracorporeal Shock Wave Therapy for Chronic Coccydynia. Medical records of 34 patients (29 females, 5 males) who had been treated with ESWT between 2017 and 2018 for chronic coccydynia were evaluated. Visual analog scale (VAS) scores were noted at the initial consultation, at each session, and during the initial and follow-up (at 6 months) examinations after the treatment. This study concluded that ESWT provided effective pain control .

In 2020, conducted a Randomized Clinical Trial on the Effect of Biofeedback on Pain and Quality of Life of Patients with Chronic Coccydynia. In this study 30 women were randomized into two groups. Both groups were injected with the corticosteroid. One group received pelvic floor muscle exercises plus biofeedback while the other group only performed exercises. The patient's pain was measured using the Visual Analog Scale (VAS) in the first visit and after 1, 2, and 6 months of follow-up as well as Dallas pain and SF-36 quality of life questionnaires before and 2 months after the treatment. This study concluded that adding biofeedback to pelvic floor muscle exercises did not lead to any further improvement in the management of chronic coccydynia .

In the 2020 aimed to evaluate the effectiveness of transrectal osteopathic manipulative treatment (OMT) for coccydynia and associated headaches. The study involved a 20-year-old female with chronic coccydynia and headaches unresponsive to conventional treatments. Following a fall and subsequent injuries during cheerleading, the patient experienced persistent pain despite various therapies. The transrectal OMT provided immediate and substantial relief in pain and associated symptoms, which was sustained over a follow-up period of 26 months. This case highlights the potential efficacy of transrectal OMT for coccydynia and suggests the need for further research on this treatment approach.

In 2018,treated 21 patients with combination therapy (Group 1) and 23 with steroid injection alone (Group 2) in a trial comparing manual therapy with steroid injection versus single steroid injection for persistent coccydynia. With a mean follow-up period of 27.8 months, the average age at the time of treatments was 30.5 years. VAS scores dropped in both groups, but the combination therapy group's outcomes were noticeably better. Just 17.4% of Group 2 experienced complete pain alleviation, compared to 61.9% of Group 1. Furthermore, whereas Group 2 experienced 73.9% of reduced VAS scores but continued discomfort, only 23.8% of Group 1 experienced this. Group 2 had a relapse rate of 56.5%, while Group 1 had no relapses. The results were unaffected by variables including the underlying etiology, BMI, coccyx morphology, or length of symptoms.

Limited number of studies have been conducted regarding coccygeal mobilization in females with coccydynia .Various methods of treating coccydynia are found in the literature but to our knowledge no research has been performed that compared the effectiveness of these interventions. Due to low levels of evidence in the published studies,additional research is needed regarding the treatment for this painful condition.

ELIGIBILITY:
Inclusion Criteria:

* Patient with coccygeal pain for more than 3 months
* Diagnosed patients of Coccydynia.
* Pain from the pericoccygeal soft tissues
* Pelvic floor muscle spasm, referred pain from lumbar pathology.

Exclusion Criteria:

* Patient with local infection (inflammatory bowel disease or psoriasis)
* Patient who undergone cocygectomy, sacroccygeal joint fusion, bleeding disorder and pregnancy.
* Spinal surgery
* Fracture of coccyx
* Having any psychological issue

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Paris Scale Questionnaire | 4th week
  The Paris Questionnaire was specifically designed for coccydynia. It covers, specifically, the functional aspects of the pain, which are not assessed by the other two questionnaires. It explores the pain when sitting (and differs, in this respect, from the VAS, which only measures the intensity of the pain), when passing from sitting to standing (very specific of coccydynia with radiologic findings), when walking and at night (pain on these occasions is frequent in severe coccydynia), and when traveling (the most sensitive detector of coccygeal pain). This set of three questionnaires offers a correct representation of the pain impact in chronic coccydynia.
DALLAS Pain Questionnaire | 4th week
  The Dallas Pain Questionnaire (DPQ), which is a 16-item visual analog tool was developed by Lawlis, McCoy, and Selby (appendix) for the purpose of evaluating subject's cognitions about the percentage that chronic pain affects four aspects of the patients' lives: 1) daily activities including pain and intensity, personal care, lifting, walking, sitting, standing, and sleeping; 2) work and leisure activities including social life, travelling, and vocational; 3) anxiety-depression and 4) social interest that includes interpersonal relationship, social support, and punishing responses.
  Each question asks the responder to rate their experience with different activities using a percentage scale from 0% to 100%. Retest reliability of DALLAS Pain Questionnaire is 0.970.
SF-36 Questionnaire in Urdu version | 4th week
  The SF-36-U is a 36 item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health. SF-36-U presented good to excellent test-retest reliability for all eight domains (ICC2,1 = 0.75-0.92. Internal consistency for all domains (Cronbach's alpha = 0.73- 0.90)

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Neelam, Principal Investigator — Riphah International University
Locations (1):
- Hafizabad Road, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nathan ST, Fisher BE, Roberts CS. Coccydynia: a review of pathoanatomy, aetiology, treatment and outcome. J Bone Joint Surg Br. 2010 Dec;92(12):1622-7. doi: 10.1302/0301-620X.92B12.25486. PMID 21119164
- [Background] Alhomedha G, Citaker S, Gunaydin G, Khan F, Sezer R. Reliability and validation of Turkish version of the Dallas Pain Questionnaire. Agri. 2022 Jan;34(1):16-22. doi: 10.14744/agri.2021.24861. PMID 34988958
- [Background] Amjad F, Mohseni-Bandpei MA, Gilani SA, Ahmad A, Zaheer A. Translation, cross-cultural adaptation, and psychometric properties of the Urdu version of Rand Short Form 36-item survey (SF-36) among patients with lumbar radiculopathy. J Bodyw Mov Ther. 2022 Oct;32:176-182. doi: 10.1016/j.jbmt.2022.05.003. Epub 2022 May 18. PMID 36180146
- [Background] Mohanty PP, Pattnaik M. Effect of stretching of piriformis and iliopsoas in coccydynia. J Bodyw Mov Ther. 2017 Jul;21(3):743-746. doi: 10.1016/j.jbmt.2017.03.024. Epub 2017 Mar 29. PMID 28750995
- [Background] Lee SH, Yang M, Won HS, Kim YD. Coccydynia: anatomic origin and considerations regarding the effectiveness of injections for pain management. Korean J Pain. 2023 Jul 1;36(3):272-280. doi: 10.3344/kjp.23175. PMID 37394271
- [Background] Maigne JY, Chatellier G, Faou ML, Archambeau M. The treatment of chronic coccydynia with intrarectal manipulation: a randomized controlled study. Spine (Phila Pa 1976). 2006 Aug 15;31(18):E621-7. doi: 10.1097/01.brs.0000231895.72380.64. PMID 16915077